CLINICAL TRIAL: NCT06218719
Title: Examining Engagement Patterns: An Observational Exploration About Tardive Dyskinesia Clinical Trials
Brief Title: Studying Patterns in Patient Engagement Among Tardive Dyskinesia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 57697757
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Tardive Dyskinesia
Keywords: tardive dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The statistical analysis of the collected data aims to reveal the many factors that influence patient involvement in clinical trials. Findings will be disseminated through conferences and scholarly papers to benefit all parties participating in clinical trials.

These findings will help to shape the design of future clinical trials for people with tardive dyskinesia, as well as enhance recruiting techniques and retention rates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of tardive dyskinesia
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* No prior treatment for tardive dyskinesia

Exclusion Criteria:

* Enrolled in another research study
* Inability to provide written informed consent
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tardive dyskinesia patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a tardive dyskinesia clinical research. | 3 months
Number of tardive dyskinesia study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horiguchi J, Watanabe K, Kondo K, Iwatake A, Sakamoto H, Susuta Y, Masui H, Watanabe Y. Efficacy and safety of valbenazine in Japanese patients with tardive dyskinesia: A multicenter, randomized, double-blind, placebo-controlled study (J-KINECT). Psychiatry Clin Neurosci. 2022 Nov;76(11):560-569. doi: 10.1111/pcn.13455. Epub 2022 Sep 17. PMID 36114799
- [Background] Hauser RA, Factor SA, Marder SR, Knesevich MA, Ramirez PM, Jimenez R, Burke J, Liang GS, O'Brien CF. KINECT 3: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Trial of Valbenazine for Tardive Dyskinesia. Am J Psychiatry. 2017 May 1;174(5):476-484. doi: 10.1176/appi.ajp.2017.16091037. Epub 2017 Mar 21. PMID 28320223
- [Background] Farrar M, Lundt L, Franey E, Yonan C. Patient perspective of tardive dyskinesia: results from a social media listening study. BMC Psychiatry. 2021 Feb 15;21(1):94. doi: 10.1186/s12888-021-03074-9. PMID 33588795

DOCUMENTS (1):
  • Informed Consent Form (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT06218719/ICF_000.pdf